CLINICAL TRIAL: NCT01767480
Title: Effects and Mechanisms of Intensive Robot-Assisted Therapy in Patients With Subacute Stroke: Outcomes in Brain/Movement Reorganization, Sensorimotor and Daily Functions, and Physiological Markers.
Brief Title: Effects of Intensive Robot-assisted Therapy in Patients With Subacute Stroke
Acronym: RT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 101-3905A3
Record Dates: First submitted 2013-01-11; First posted 2013-01-14 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Stroke
Keywords: Intensive Robot Assisted Therapy; Subacute Stroke; Brain Reorganization; Sensory Motor; Physiological Marker
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Higher-intensity RT group (Experimental): All participants received a duration-matched intervention for 90-120 minutes/day, 5 days/week for 4 consecutive weeks. For the RT groups, they will receive RT training together with functional rehabilitation trainings. Within 1 training session, each patient in the higher-intensity RT group will use Bi-Manual-Tract to practice 400-600 repetitions of the mode 1 and 800-1000 repetitions of mode 2, totaling 1200-1600 repetitions, respectively for the forearm and the wrist movements. In addition, the patients will practice 100-200 repetitions in mode 3, if application.
  Interventions: Device: RT; Behavioral: Conventional rehabilitation (CR)
- Lower-intensity RT group (Experimental): Patients in the lower-intensity RT received half the number of the repetitions per unit of time than patients in the higher-intensity RT group. Within 1 training session, patients in the lower-intensity RT group will practice 200-300 repetitions of the mode 1 and 400-500 repetitions of mode 2, totaling 600-800 repetitions, respectively for the forearm and the wrist movements. In addition, the patients will practice 50-100 repetitions in mode 3, if application.
  Interventions: Device: RT; Behavioral: Conventional rehabilitation (CR)
- Conventional rehabilitation (CR) group (Active Comparator): The CR group will be designed to control for the duration of therapeutic activities. CR will focus on neurodevelopmental techniques with emphasis on functional tasks when possible. The functional training will be designed based on patients' motor capacity and include gross motor and fine motor dexterity training, and transitive and intransitive training. Stretching of the more affected limb, passive and active range of movements, and normalizing muscle tone by applying reflex inhibition patterns, inhibiting abnormal patterns, weight bearing with the affected limb will be applied to assist in functional task practice.
  Interventions: Behavioral: Conventional rehabilitation (CR)

INTERVENTIONS:
Device: RT — The Bi-Manu-Track enables the symmetrical practice of 2 movement patterns in conjunction with computer games: forearm pronation-supination and wrist flexion-extension. Each movement has three computer-controlled modes: (1) passive-passive, with both arms being moved by the machine with speed and range of motion individually adjustable; (2) active-passive, with the nonaffected arm driving the affected arm in a mirror-like fashion; and (3) active-active, with both arms actively moving against resistance. The speed of movement, the amount of resistance, and the range of movement can be adjusted individually. The device has a mechanical breaking of the movement when the torques exceeded 4 Nm, emergency breaks in the reach of the patients, skin friendly materials, and minimal risk for contusions.
  Other Names: Bi-Manu-Track; Reha-Stim Co., Berlin, Germany
  Arms: Higher-intensity RT group; Lower-intensity RT group
Behavioral: Conventional rehabilitation (CR) — CR will focus on neurodevelopmental techniques with emphasis on functional tasks when possible. The functional training will be designed based on patients' motor capacity and include gross motor and fine motor dexterity training, and transitive and intransitive training. Stretching of the more affected limb, passive and active range of movements, and normalizing muscle tone by applying reflex inhibition patterns, inhibiting abnormal patterns, weight bearing with the affected limb will be applied to assist in functional task practice.
  Other Names: CR

SUMMARY:
Robot-assisted training (RT) devices developed to date have a significant impact on stroke rehabilitation. Several research groups have developed the robotic devices and examined their efficacy on improving upper limb function after stroke. All these robotic devices have been applied in stroke rehabilitation and their efficacy are evaluated, but the scientific evidence for the mechanisms of RT-induced recovery, the optimal treatment intensity, and the impact on physiological responses is still lacking.

This trial is to examine (1) the immediate effects of treatment intensity in RT on sensorimotor impairments and functional performance in patients with subacute stroke; (2) the long-term benefits of treatment intensity in RT by conducting a 6-month follow up evaluation; and (3) the effects of RT on cortical/movement reorganization as well as on the physiological markers of inflammation, oxidative stress, and erythrocyte deformability. These overall findings will help better understanding of the efficacy of RT on functional outcomes, brain and movement reorganization, and physiological markers.

DETAILED DESCRIPTION:
Subacute stroke participants will be recruited from the Chang Gung Memorial Hospital and then were randomly assigned to 1 of the 3 groups: RT with higher-intensity group, RT with lower-intensity group, and conventional intervention group. Assessments on sensorimotor impairments (Fugl Mayer Assessment, Motor Status Scale, Modified Ashworth Scale, Myoton, Muscle Metabolism, Box and Block Test, and Revised Nottingham Sensory assessment) and functional performance (Functional Independence Measure, Motor Activity Log, ABILHAND Questionnaire, Adelaide Activities Profile, EQ-5D-5L, and accelerometer) take about 40 minutes to complete. Evaluation of brain reorganization using functional magnetic resonance image and movement patterns by kinematic analysis take about 1 hour for each examination. Blood samples of the patients (12 ml.) will be collected to examine the physiological markers (ie, inflammation-related markers, oxidative stress markers, and erythrocyte deformability) before and after intervention. Total 24 ml blood will be collected in this study. Except for the blood taking, all the examinations are non-invasive.

ELIGIBILITY:
Inclusion Criteria:

* first episode of unilateral stroke
* time since stroke less than 3 months, i.e., acute or subacute stage
* initial motor part of upper limb of FMA score ranging from 10 to 40, indicating severe to moderate movement impairment
* no serious cognitive impairment (i.e., Mini Mental State Exam score > 23)

Exclusion Criteria:

* pregnant or breastfeeding women
* aphasia that might interfere with understanding instructions
* major health problems or poor physical conditions that might limit participation
* currently participation in any other research. Potential participants will be also excluded if they have any contraindication to fMRI scanning including claustrophobia, seizures, the presence of pacemaker, mental elements (e.g., steel nails) inside the body or in the eyes, and excessive obesity.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-01; Primary Completion 2015-02 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment (FMA) | At baseline and immediately after the completion of intervention
  The upper limb part of FMA will be used to evaluate sensorimotor impairment. The motor part consists of 33 items for the reflexes and movement of shoulder, elbow, forearm, wrist, hand, and coordination/speed. The non-motor part consists of 30 items for sensation, passive joint motion, and joint pain of the upper limb. Each item is scored on a scale of 0-2 with a maximum of 66 for motor part and 60 for non-motor (sensory) part. Higher score indicates better sensorimotor function of upper limb.
Motor Status Scale (MSS) | At baseline and immediately after the completion of intervention
  The MSS will be used to identify and quantify change of motor function of upper limb after stroke. This scale isolates and grades movement of the shoulder, elbow, forearm, and wrist using a 6-point scale (0, -1, 1, +1, -2, 2), ranging from no volitional movement to faultless movement. Scoring for the hand is based on a 3-point scale (0-2). It consists of 2 subscales including shoulder/elbow scale and wrist/finger scale. The subscale of shoulder/elbow scale consists of the sum of measures of 12 shoulder movements and 5 elbow/forearm movements (maximum score = 40). The subscale of wrist/finger consists of the sum for 3 wrist and 15 hand movements and 3 hand-based functional tasks (maximal score = 42).
Modified Ashworth Scale (MAS) | At baseline and immediately after the completion of intervention
  The MAS is the most frequently used clinical rating scale to measure muscle spasticity. This measure involves manually moving a limb through the range of motion (ROM) to passively stretch specific muscle groups. The grades of spasticity in MAS are as follows: 0=No increase in muscle tone; 1=Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is(are) moved in flexion or extension; 1+=Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM; 2=More marked increase in muscle tone through most of the ROM, but affected part(s) easily moved; 3=Considerable increase in muscle tone, passive movement difficult; 4=Affected part(s) rigid in flexion or extension.
MyotonPRO | At baseline and immediately after the completion of intervention
  The Myoton is a hand-held device measure of three mechanical properties of muscle: tone, stiffness and elasticity. Three measurement parameters in the Myoton: F - Frequency, Hz, characterizes muscle tone; D - Decrement, characterizes muscle elasticity; S - Stiffness, N/m, characterizes muscle stiffness. There have been several prototypes of Myoton. Present study will use MyotonPRO; the basic principle is the same in all prototypes but the MyotonPRO has several updates such as a triaxial accelerometer. Comparing with the single axis accelerometer in the earlier prototypes, MyotonPRO makes it more feasible for application.
Muscle metabolism (NIRS) | At baseline and immediately after the completion of intervention
  Muscle metabolic dysfunction will be measured by the near-infrared ray spectroscopy (NIRS). The NIRS will be applied to both the affected and the unaffected arms. The NIRS sensor will be fixed on the targeted muscle of one of the forearms and a cuff is placed on the upper arm of the same side. The artery occlusion will be applied by inflating the cuff to a pressure of at least 60 to 80 above systolic pressure to block both venous outflow and artery inflow. The artery occlusion will last approximate 30 seconds then the cuff pressure is released. The decrease rate of oxyhemoglobin and the increase rate of deoxyhemoglobin during artery occlusion can reflect muscle's anaerobic metabolism during vasoconstriction. The hyperaemic response of the muscle during recovery phase can be characterized by reoxygenation rate and recovery time.
Box and Block Test (BBT) | At baseline and immediately after the completion of intervention
  The BBT will be used as a test of manual dexterity. There are 150 blocks in a test box. When testing begins, the subject should grasp one block at a time with dominant hand, transport the block over the partition, and release it into the opposite compartment. Instruction of this test is "I want to see how quickly you can pick up one block at a time with your right (or left) hand [point to the hand]. Carry it to the other side of the box and drop it. Make sure your fingertips cross the partition." The testing time is one minute. Then, the procedure will be repeated with the nondominant hand. After testing, the examiner should count the blocks. The score is the number of blocks carried from one compartment to the other in one minute. Score for each hand will be separately calculated.
Revised Nottingham Sensory Assessment (RNSA) | At baseline and immediately after the completion of intervention
  The changes on somatosensory function will be determined by the RNSA. This is a standardized tool with good reliability to measure sensory function in the stroke population.The RNSA includes 3 major types of sensation: tactile sensation, proprioception, and stereognostic sense. For the purpose of this study, the regions of upper limb will be selected to be assessed.
Functional Independence Measure (FIM) | At baseline and immediately after the completion of intervention
  The FIM consists of 18 items grouped into 6 subscales measuring self-care, sphincter control, transfer, locomotion, communication, and social cognition ability. Each item is rated from 1 to 7 (maximum score 126) based on the required level of assistance to perform the tasks (e.g., 1-complete assistance and 7-complete independence). A low score on any subscale indicates a more severe disability.
Motor Activity Log (MAL) | At baseline, immediately after the completion of intervention, at a 6-month follow up
  The MAL will be used to capture the level of use of affected upper limb in daily living. The MAL is a semi-structured interview assessing the amount of use (AOU) and quality of movement (QOM) of the affected arm in 30 main daily activities. It scores 0-5 for each activity. Higher score means better performance of the affected arm.
ABILHAND Questionnaire | At baseline, immediately after the completion of intervention, at a 6-month follow up
  The ABILHAND Questionnaire will be used to evaluate the ability of upper limb in bimanual activities. There are 23 bimanual activities to measure subjectively perceived difficulty of patients in performing some common activities in daily living, such as buttoning, cutting nails, and opening a bottle. It scores on a scale of 0-3 (0-cannot perform, 1-performs partially or with great difficulty, 2-performs with some difficulty, 3-performs fully). Its reliability and construct validity has been confirmed.
Adelaide Activities Profile (AAP) | At baseline, immediately after the completion of intervention, at a 6-month follow up
  The AAP will be applied to indicate the level of participation in household and community activities. This profile includes 21 activities in the four areas: domestic chores, household maintenance, service to others, and social activities. It scores on a scale of 0-3, with higher score indicating more frequent participation.
EQ-5D-5L | At baseline and immediately after the completion of intervention
  The EQ-5D-5L is an instrument for measuring health status. It consists of the descriptive system and the EQ visual Analogue scale (EQ VAS). The descriptive system comprises the same 5 dimensions (mobility, self care, usual activities, pain/discomfort, and anxiety/depression). There are 5 levels for each dimension: no problems, slight problems, moderate problems, severe problems, and extreme problems. The EQ VAS records the respondent's self-rated health on a 20 cm vertical, visual analogue scale with endpoints labeled 'the best health you can imagine' and 'the worst health you can imagine'.
Accelerometers | At baseline, immediately after the completion of intervention, at a 6-month follow-up.
  The activity monitors (i.e. accelerometers) will be used to provide a direct and objective measure of the amount of the impaired arm movement outside the laboratory. This measure, quantitatively recording the amount of activity in free-living conditions, will be used to reflect increase in the amount of affected arm use over time. The participants will be asked to wear an accelerometer on each arm for 3 consecutive days to measure what they actually do. The accelerometers to be used will be wireless plastic units about the size and weight of a large wristwatch that will be worn proximal to the wrist on terrycloth bands.
Functional magnetic resonance imaging (fMRI) | At baseline and immediately after the completion of intervention
  Participants will receive fMRI scanning before and after the intervention on a 3T clinical MRI scanner at Chang Gung Memorial Hospital in Linkou. During the scanning sessions, the head and the unaffected hand of the participants will be restrained and stabilized in a head coil and by a customized splint mask and a wooden apparatus with straps, respectively. Both of their upper limbs will be posited by their torsos. During the two sessions of examination, the relative activity time courses of the blood oxygenation level-dependent (BOLD) response will be collected for further analysis.
Kinematic analysis | At baseline and immediately after the completion of intervention
  The kinematic analysis will involve unilateral and bilateral tasks, in which the participants will be asked to perform by using the affected upper limb or both upper limb simultaneously. A motion analysis system with 7 cameras (VICON MX 30d, Oxford Metrics Inc., Oxford, UK) will be used to capture the motion of arm (s) in kinematic testing. The markers will be attached on the styloid processes of the ulna. Depending on the unilateral or bilateral tasks, the makers will be placed on the affected arm or the both arms, respectively.
Inflammatory markers | At baseline and immediately after the completion of intervention
  Proinflammatory markers and anti-inflammatory markers will be used to reflect the changes on inflammation. Proinflammatory markers include C-reactive protein, tumor necrosis factor-α (TNF-α), interleukin (IL)-1β, IL-6, soluble intercellular adhesion molecule (sICAM), and matrix metalloproteinase 9 (MMP 9). Anti-inflammatory markers include IL-10 and IL-1 receptor antagonist.
Oxidative stress markers | At baseline and immediately after the completion of intervention
  Oxidative stress markers and antioxidative markers will be used to reflect the changes on oxidative stress. Oxidative stress makers include malondialdehyde (MDA), 8-Hydroxy-2-deoxyguanosine (8-OHdG), and immunoglobulin G (IgG), whereas antioxidants include superoxide dismutase (SOD), glutathione peroxidase (GPx), and catalase.
Erythrocyte deformability | At baseline and immediately after the completion of intervention
  The Elongation Index (EI) will be used to determine the red blood cell deformability, which is based on an isointensity curve in the diffraction pattern by using an ellipse-fitting program. EI is calculated by (L-W)/(L+W), where L and W are the major and minor axes of the ellipse, respectively. The deformability index (δ) is defined as the ratio of the major to the minor axis length (L/W).
Blood glucose indicators | At baseline and immediately after the completion of intervention
  To investigate the relationships between blood glucose levels and functional outcomes, we will also test the level of glucose and HbA1C for the participants before and after rehabilitation intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Yi Wu, ScD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Kwei-Shan, Tao-Yuan, Taiwan

REFERENCES:
- [Derived] Clark B, Whitall J, Kwakkel G, Mehrholz J, Ewings S, Burridge J. The effect of time spent in rehabilitation on activity limitation and impairment after stroke. Cochrane Database Syst Rev. 2021 Oct 25;10(10):CD012612. doi: 10.1002/14651858.CD012612.pub2. PMID 34695300